CLINICAL TRIAL: NCT03939442
Title: Evaluation of Patients Who Underwent Sleeve Gastrectomy With Jejunoileal Anastomosis for the Treatment of Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, cihan gokler, Inonu, Inonu University
Other Study IDs: 2019/3-10
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-05

CONDITIONS: Sleeve Gastrectomy With Jejunoileal Anastomosis
Keywords: obesity, diabetes mellitus, bariatric surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sleeve gastrectomy with jejunoileal anastomosis — The sleeve gastrectomy was performed first, after using a sealer and divider device to dissect the omentum away from the greater gastric curvature from approximately 5 cm proximal to the pylorus up to the angle of His. Excision of the fundus and the body of the stomach was then performed with a laparoscopic linear stapler upon a 36 French orogastric tube (bougie). An isoperistaltic side-to-side anastomosis between the jejunum (at 50 cm distal to the Treitz ligament) and the distal ileum ( at 200 cm proximal to the ileocecal valve) was then created using the same linear stapler with a blue cartridge (3.5 mm). A soft Penrose drain was left at the subdiaphragmatic space, and the abdominal wound was closed.

SUMMARY:
Laparoscopic sleeve gastrectomy operations performed for morbid obesity are among the most common methods in the world. Gastric or intestinal bypass surgery with or without sleeve gastrectomy is thought to be more effective in controlling both weight loss and metabolic diseases. For this purpose, Roux-en-y gastric bypass, transit bipartition, duodenal switch, jejunoileal bypass are performed. The aim of this study was to evaluate the effects of jejunoileal bypass surgery on weight loss and metabolic diseases in patients with sleeve gastrectomy.

DETAILED DESCRIPTION:
Bariatric surgery results in more and more long-term weight loss than traditional treatment in moderate and severe obesity. Due to morbid obesity, jejunoileal bypass has been applied since 1970. Laparoscopic sleeve gastrectomy and jejunoileal anastomosis are among the rare techniques described in 2012. There are few studies on this technique.

Between 2015 and 2018, jejunoileal bypass operations with laparoscopic sleeve gastrectomy for morbid obesity will be evaluated in Inonu University gastroenterology surgery clinic. The patients' age, gender, body mass index, weight loss in follow-up periods, whether there is back weight gain, the effects on metabolic diseases, early and late complications will be evaluated.

ELIGIBILITY:
Inclusion Criteria:All patients who underwent the sleeve gastrectomy with jejunoileal bypass between 2015-2018 for the treatment morbid obesity

Exclusion Criteria:other operations for morbid obesity except sleeve gastrectomy with jejunoileal bypass

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged between 18 and 60 years with a body mass index greater than 40, no comorbidity or a body mass index of 35-40, with a comorbidity (diabetes mellitus, hypertension, obstructive sleep apnea)
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Excess weight loss | 2 years
  body mass index (BMI) 25 was considered ideal. The ratio of the value above this value to the value that arrived at the end of 2 years was calculated. Over 80% was considered successful.
diabetes remission | 2 years
  1. Complete remission absence antidiabetic medications, HbA1c level below 6%, fasting blood glucose value below 100 mg / dl
  2. partial remission Subdiabetic hyperglycemia (HbA1c 6%-6.4%, FBG 100-125 mg/dL) in the absence antidiabetic medications
  3. Unchanged The absence of remission or improvement as described earlier

CONTACTS AND LOCATIONS:
Locations (1):
- Cihan Gökler, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided